CLINICAL TRIAL: NCT04623671
Title: A Randomized, Double-Blind, Placebo-Controlled Study Evaluating the Safety and Efficacy of Intravenous Infusion of CAP-1002 in Patients With COVID-19 (INSPIRE)
Brief Title: Intravenous Infusion of CAP-1002 in Patients With COVID-19
Acronym: INSPIRE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Capricor Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAP-1002-COVID-19-02
Record Dates: First submitted 2020-10-07; First posted 2020-11-10 (Actual); Results first posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Covid19
Keywords: SARS-CoV-2; COVID; COVID-19; COVID19
MeSH Terms: conditions — COVID-19 | interventions — chenodeoxycholate sulfate conjugate

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Syringes (60-mL) with amber film-covered barrels
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CAP-1002 (Active Comparator): The active pharmaceutical ingredient in CAP-1002 is Cardiosphere-Derived Cells (CDCs). CDCs are known to secrete numerous bioactive elements (growth factors, exosomes) which impact the therapeutic benefits of the cell-based therapy. The mechanism of action is the composite ability to be immunomodulatory, anti-fibrotic, anti-inflammatory, and pro-angiogenic.
  Interventions: Biological: CAP-1002
- Placebo (Placebo Comparator): Matching placebo solution
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CAP-1002 — Peripheral infusion of 150 million cardiosphere-derived cells (CDCs)
  Other Names: Allogeneic Cardiosphere-Derived Cells; CDCs
  Arms: CAP-1002
Biological: Placebo — Matching placebo solution
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, Pilot, Phase 2 Exploratory study that will enroll subjects with a clinical diagnosis of COVID-19 confirmed by laboratory testing and who are in severe or critical condition as indicated by life-support measures.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled Pilot, Phase 2 Exploratory study that will enroll subjects with a clinical diagnosis of COVID-19 confirmed by laboratory testing and who are in severe or critical condition as indicated by life-support measures. Prior to protocol procedures, informed consent will be obtained from the subject or a legally authorized representative. Subjects will undergo a screening evaluation to determine eligibility based on the protocol inclusion and exclusion criteria.

The primary objectives of the study are to determine the safety and effectiveness of intravenously infused CAP-1002 in improving clinical outcomes in severely or critically ill patients with COVID-19.

Eligible subjects will be randomized to either the CAP-1002 or placebo group (1:1 ratio) and undergo baseline safety and efficacy assessments approximately 1 to 5 days prior to the administration of investigational product (IP). Treatment administration consists of IP consisting of 150M CDCs or matching placebo on study Day 1. Background standard of care treatment and practices will be maintained for all patients enrolled in the study.

Subjects will complete Screening followed by a Treatment and Follow-up phase. A detailed medical history will be collected, including the presence of any co-morbidities and risk factors believed to be associated with COVID-19 outcomes or emergent factors since the time of infection. Eligibility must be reviewed and confirmed on Day 1 prior to the infusion of IP.

Subjects will be observed during the index hospitalization and monitored for outcome and safety with vital signs (heart rate, blood pressure, respiratory rate, and oxygen saturation), physical examinations, electrocardiograms, clinical laboratory testing including complete blood count and comprehensive metabolic panel, inflammatory markers and adverse events. Blood samples will be collected and submitted to a central laboratory for future proteomic assay assessment. Use of any concomitant medications to treat COVID-19 will be documented.

Follow-up will be conducted on Days 2, 3, 7, 15, 30, 60, and 90 either in the inpatient setting or by telephone if the subject has been discharged. All subject participation will be a maximum of 13 weeks from Screening.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects at least 18 years of age at time of consent.
2. Diagnosis of SARS-CoV-2 infection confirmed by real-time reverse transcription polymerase chain reaction (RT-PCR) assay.
3. Compromised respiratory status as defined by arterial oxygen saturation < 92% (oxygen saturation measured by pulse oximetry) OR cardiomyopathy due to COVID-19 (defined as a new drop in ejection fraction to ≤ 50% during COVID-19 with no evidence of obstructive coronary artery disease based on medical records review).
4. Elevation of at least 1 inflammatory marker (IL-1, IL-6, IL-10, TNF-α, ferritin, CRP) defined as ≥ 2x upper limit of laboratory normal reference value.
5. Written informed consent provided by subject or legal representative.

Exclusion Criteria:

1. Currently receiving extracorporeal membrane oxygenation (ECMO) or high frequency oscillatory ventilation (HFOV).
2. Patients who have been intubated.
3. Patients with established positive bacterial blood cultures prior to enrollment or suspicion of superimposed bacterial pneumonia.
4. Patients with untreated human immunodeficiency virus (HIV) infection.
5. Creatinine clearance less than 30 mL/minute.
6. Liver function tests > 5x normal.
7. Current or history (within the previous 5 years) of systemic autoimmune or connective tissue disease.
8. Known allergy or hypersensitivity to any of the IP constituents such as dimethyl sulfoxide (DMSO) or bovine proteins.
9. Treatment with a cell therapy product within 12 months prior to randomization.
10. Participation in an ongoing protocol studying an experimental drug or device.
11. Pregnant or breastfeeding female subjects, and sexually active female subjects of childbearing potential not willing to use contraceptive methods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2020-11-15 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Albertson, MD, Principal Investigator — UC Davis
Locations (4):
- United States (4):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California Davis, Sacramento, California
  - Henry Ford Health System, Detroit, Michigan
  - PharmaTex Research, LLC, Amarillo, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CAP-1002: Participants received 1 peripheral IV infusion of IP (2 × 75M for a total of 150M CDCs administered at the clinical site).
- Placebo: Participants received 1 infusion of intervention matching placebo on Day 1.
Period: Overall Study
Arm/Group | CAP-1002 | Placebo
Started | 28 | 27
Completed | 21 | 20
Not Completed | 7 | 7
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 2 | 1
Not completed — Death | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CAP-1002 | Placebo | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (14.13) | 55.0 (11.6) | 56.4 (12.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 7 | 21
  Male | 14 | 20 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 22
  Not Hispanic or Latino | 16 | 15 | 31
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 22 | 18 | 40
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety of CAP-1002: Incidence of All-Cause Mortality
Description: Number of all-cause mortality cases from start of treatment up to end of study. Survival was measured as the time between the date of the start of treatment and the date of death.
Time Frame: Up to End of Study (Day 90)
Population: Safety analysis set includes all enrolled participants who were randomized and received at least 1 dose of randomized investigational product, CAP-1002 or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | CAP-1002 | Placebo
Number analyzed (Participants) | 28 | 27
Participants | 5 | 6

ADVERSE EVENTS:
Time Frame: Up to end of study (Day 90).
Description: Safety analysis set includes all enrolled participants who were randomized and received at least 1 dose of randomized investigational product, CAP-1002 or placebo.
Arm/Group | CAP-1002 | Placebo
All-Cause Mortality (participants affected / at risk) | 5/28 | 6/27
Serious Adverse Events (participants affected / at risk) | 9/28 | 7/27
Other Adverse Events (participants affected / at risk) | 21/28 | 16/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAP-1002 (N=28) | Placebo (N=27)
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Covid-19 (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia pseudomonal (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 2 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Acute respiratory distress failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Tachypnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CAP-1002 (N=28) | Placebo (N=27)
Anaemia (Blood and lymphatic system disorders) | 2 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 2
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 3
Atrial flutter (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1
Chronic left ventricular failure (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Left ventricle outflow tract obstruction (Congenital, familial and genetic disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Anorectal discomfort (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 0 | 1
Hypothermia (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 1
Pyrexia (General disorders) | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 1 | 0
Aspergillus infection (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1
Bacterial infection (Infections and infestations) | 0 | 1
Balanitis candida (Infections and infestations) | 1 | 0
Candida infection (Infections and infestations) | 2 | 0
Cytomegalovirus oesophagitis (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 0 | 1
Oesophageal candidiasis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 1
Sepsis syndrome (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 2 | 4
Serratia infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Urinary tract infection fungal (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis; Aspergillus infection (Infections and infestations) | 1 | 0
Tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Cryptococcus test positive (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Inflammatory marker increased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Spasmodic dysphonia (Nervous system disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 1 | 4
Azotaemia (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 1
Hypertension (Vascular disorders) | 1 | 0
Hypertensive urgency (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 4 | 2
Ischaemia (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-03-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT04623671/Prot_000.pdf
  • Statistical Analysis Plan (2022-02-26): https://cdn.clinicaltrials.gov/large-docs/71/NCT04623671/SAP_001.pdf